CLINICAL TRIAL: NCT03513510
Title: Participatory Development and Pilot Testing of iChoose: An Adaptation of an Evidence-Based Pediatric Weight Management Program for Community Implementation
Brief Title: Development and Pilot Testing of a Childhood Obesity Treatment Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Pittsylvania/Danville Health District (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Children's Healthcare Center (Unknown); Boys and Girls Club of Danville (Unknown); Danville Parks and Recreation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VT IRB 12-977; R24MD008005 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2019-02

CONDITIONS: Childhood Obesity
Keywords: evidence-based programs; community-based participatory research; program adoption
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iChoose (Experimental): 6 biweekly family sessions, 6 biweekly telephone support calls to parents, 6 biweekly newsletters for children, and 3 supervised exercise sessions per week/3 months; delivers intervention to parents and children only
  Interventions: Behavioral: iChoose

INTERVENTIONS:
Behavioral: iChoose

SUMMARY:
The primary aims were to assess community capacity to develop, implement, and sustain a childhood obesity reduction initiative in the health-disparate Dan River Region as well as to pilot test iChoose to determine the potential reach (i.e., proportion of target population & representativeness), effectiveness (i.e., changes in child BMI z-scores over a 6 month period), feasibility (i.e., the degree to which the intervention can be adopted, implemented, and sustained as intended) and cost (i.e., resource and staffing costs) of the newly developed intervention.

DETAILED DESCRIPTION:
The Dan River Region (DRR) is a federally designated medically under-served area/population with high rates of obesity. In response to 3 comprehensive community needs assessments The Dan River Partnership for a Healthy Community (DRPHC) was established in 2010 'to foster community partnership to combat obesity in the Dan River Region through healthy lifestyle initiatives' (DRPHC mission statement). To date the DRPHC (1) tested a successful adult weight control intervention, (2) initiated youth-focus community garden and instant recess initiatives, and (3) continues to complete a comprehensive audit of the food and physical activity environment across the DRR. This RFA provided an opportunity to address an additional and complimentary area of need for the DRPHC-childhood obesity. A newly formed subcommittee and community advisory board (CAB) of the DRPHC, Partnering for Obesity Planning and Sustainability (POPS), met in preparation of this proposal and discussed the need to engage systems where high need families received services and could participate in childhood obesity treatment. The POPS-CAB came to consensus that using a systems-based approach, within the existing CBPR partnership would allow for the development of a contextually relevant intervention with the potential for long-term sustainability. Systems-based approaches include, but also move beyond, a focus on initiative effectiveness and address broader contextual issues such as initiative adoption, implementation, and maintenance across settings and delivery staff as well as reach and maintenance of effects at the individual level. The general goal of this proposal is to engage multiple systems through the DRPHC POPS-CAB and design and test prototype childhood obesity interventions. The current membership of the POPS-CAB include Danville Pittsylvania Health District, Children's Healthcare Center, Danville Parks Recreation & Tourism, and Boys & Girls Club, along with an interdisciplinary team of academic investigators. The first aim is to assess community capacity to develop, implement, and sustain a childhood obesity reduction initiative in the DRR. To accomplish this aim a concurrent mixed-method study design will be used and guided dimensions of community capacity and organizational level dimensions of the RE-AIM framework (i.e., adoption, implementation, and maintenance). The second aim is to determine the potential reach, effectiveness, feasibility and cost of the newly developed interventions. Three stages of iterative intervention testing/formative feedback loops in a public health and healthcare system will be used to achieve this aim. The partnership members will meet in an ongoing basis to discuss the qualitative & quantitative results and make adaptations to improve the strategies. Indicators of success include reduced child BMI z-scores, the engagement of multiple systems, and regional capacity to evaluate research evidence and integrate this evidence into sustainable practices. The end goal is a childhood obesity intervention that is ready for large scale testing across these systems in the DRR.

ELIGIBILITY:
Inclusion Criteria:

* Parent/child dyads were eligible for participation if they resided in the Dan River Region
* English speaking
* child with a BMI percentile ranking of 85 or higher

Exclusion Criteria:

* children with a major cognitive impairment and parents or children with a medical contraindication for moderate physical activity

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-06-27 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Community capacity to identify, adapt, and implement a childhood obesity program. | 2 years
  qualitative interviews

SECONDARY OUTCOMES:
child BMI z-score | 6-months
  This is a age and gender normed standardization of child weight status.
reach | 6-months
  the proportion of eligible families that enroll in the trial and their representativeness to the larger population of eligible families.
cost | 6 months
  cost of intervention delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Estabrooks, PhD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No
There is no current plan. Though we will comply with requests consistent with NIH data sharing policies.